CLINICAL TRIAL: NCT01993992
Title: Parental Anxiety and Its Relationship With Pediatric Patients' Post-operative Responses
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310021RIND
Record Dates: First submitted 2013-11-03; First posted 2013-11-25 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Post-operative Delirium; Children; Anxiety
Keywords: Anesthesia
MeSH Terms: conditions — Emergence Delirium; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-operative delirium had multiple risk factors, such as pre-operative anxiety status, post-operative pain, and anesthetic method. We currently decrease pre-operative anxiety by parental accompanying until the children put to sleep. However, references indicate that parental anxiety can increase the post-operative delirium. Heart rate variability was used to measure the anxiety status of parents. We think sympathetic tone elevation measured by heart rate variability may not induce by anxiety alone, thus we want to explore this question by using Stat-Trait Anxiety Inventory questionnaire.

DETAILED DESCRIPTION:
Outcome measures

1. Post-operative emergence delirium, observed with an average duration up to 24 hours
2. Sedatives used in recovery unit

ELIGIBILITY:
Inclusion criteria:

* American Society Anesthesia (ASA) risks classification I or II

Exclusion criteria:

* Parents who have cognitive problems
* Parents who have difficulty finishing questionnaire

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Age younger than 16-year-old who required surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
degree of emergence delirium | after operation, with an average duration up to 24 hours

SECONDARY OUTCOMES:
recovery room stay time | after operation, with an average duration up to 24 hours
Sedatives used in recovery room | after operation, with an average duration up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: YI-CHIA WANG, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan